CLINICAL TRIAL: NCT05790499
Title: Continuous Atorvastatin Therapy Compared With Intermittent Atorvastatin Therapy for the Effect of LDL-c Level Variability and the Regulation of Trained Immunity
Brief Title: LDL-c Level Variability and Trained Immunity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiang Cheng, professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Atorvastatin-007
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Cholesterol Variability; Trained Immunity
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atorvastatin (Experimental)
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Patients are treated with atorvastatin for 2 weeks (40 mg/day), atorvastatin free for 2 weeks, atorvastatin treatment for 2 weeks, atorvastatin free for 2 weeks, a 4-week washout period (no treatment), and atorvastatin treatment for the last 4 weeks.

SUMMARY:
Statin treatment significantly reduces the incidence of cardiovascular events. However, cholesterol variability is associated with the risk of adverse events such as mortality, myocardial infarction, and stroke. The previous research found that the inflammatory activity of peripheral blood mononuclear cells in mice fed with intermittent high-fat diet was significantly increased, and the cholesterol variability had an impact on the trained immunity of peripheral blood mononuclear cells, thus aggravating the atherosclerosis in mice.

We plan to compare the differences in serum LDL-C levels after intermittent atorvastatin treatment and continuous atorvastatin treatment, and investigate the impact of this difference on the trained immunity of peripheral blood mononuclear cells.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate, understand and sign an informed consent form;
2. Age ≥ 18 years old, male or postmenopausal female (defined as amenorrhea over 2 years with relevant clinical characteristics, such as age over 55 years old or menopausal cardiovascular symptoms such as hot flashes, night sweats, palpitations, etc.). Women with hysterectomy and/or bilateral oophorectomy may also be considered for inclusion in the group;
3. Commit to complying with research procedures and cooperate in the implementation of the entire process of research; 4、LDL-c>3.4mmol/L

Exclusion Criteria:

1. Previous cardiovascular history;
2. Statins should not be discontinued in high-risk groups for cardiovascular events;
3. Any known organ dysfunction;
4. Intolerance to statins;
5. Pregnant women, lactating women, or women of childbearing age who do not use effective contraception;
6. Participating in other clinical trials;
7. Unable to follow the study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes in LDL-C levels between baseline and atorvastatin treatment cycles | 16 weeks
  in the phase of atorvastatin intermittent treatment and continuous treatment

SECONDARY OUTCOMES:
PBMCs subgroup percentage and activation status | 16 weeks
  in the phase of atorvastatin intermittent treatment and continuous treatment
PBMCs secreting cytokines | 16 weeks
  in the phase of atorvastatin intermittent treatment and continuous treatment
Differences in gene expression of PBMCs | 16 weeks
  in the phase of atorvastatin intermittent treatment and continuous treatment
The levels of hs-CRP, IL-6, IL-18, and sVCAM-1 | 16 weeks
  in the phase of atorvastatin intermittent treatment and continuous treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China